CLINICAL TRIAL: NCT00662740
Title: 1-yr Study Comparing TioSal Combo Regimens Versus Single Agent Therapies (Spiriva HandiHaler and Salmeterol PE Capsule)
Brief Title: Tiotropium/Salmeterol Inhalation Powder (Spiriva Handihaler and Salmeterol Polyethylene (PE) Capsule) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.14; 2007-005134-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (5):
- Tiotropium/Salmeterol quaque die (QD, once daily) (Experimental): Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule
  Interventions: Drug: Tiotropium/Salmeterol QD
- Tiotropium quaque die (QD, once daily) (Active Comparator): Tiotropium Inhalation Powder, hard gelatine capsule (Spiriva®)
  Interventions: Drug: Tiotropium (Spiriva®)
- Salmeterol bis in die (BID, twice daily) (Active Comparator): Salmeterol Inhalation Powder, hard PE capsule
  Interventions: Drug: Salmeterol
- Tiotropium/Salmeterol quaque die (QD, once daily)+ Salmeterol (Active Comparator): Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule, plus Salmeterol Inhalation Powder, hard PE capsule
  Interventions: Drug: Tiotropium/Salmeterol QD+ Salmeterol
- Placebo (Placebo Comparator): Placebo Inhalation Powder, hard PE capsule / hard gelatine capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium/Salmeterol QD — Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule
  Arms: Tiotropium/Salmeterol quaque die (QD, once daily)
Drug: Placebo — Placebo Inhalation Powder, hard PE capsule / hard gelatine capsule
  Arms: Placebo
Drug: Salmeterol — Salmeterol Inhalation Powder, hard PE capsule
  Arms: Salmeterol bis in die (BID, twice daily)
Drug: Tiotropium/Salmeterol QD+ Salmeterol — Tiotropium/Salmeterol Inhalation Powder, Hard Polyethylene Capsule, plus Salmeterol Inhalation Powder, hard PE capsule
  Arms: Tiotropium/Salmeterol quaque die (QD, once daily)+ Salmeterol
Drug: Tiotropium (Spiriva®) — Tiotropium, Spiriva®
  Arms: Tiotropium quaque die (QD, once daily)

SUMMARY:
The primary objectives of this study are to assess bronchodilator efficacy as determined by forced expiratory volume in one second (FEV1), the effect on dyspnoea as determined by the Baseline Dyspnoea Index/Transition Dyspnoea Index (BDI/TDI), the effect on health status as determined by the St George Respiratory Questionnaire (SGRQ) and the effect on chronic obstructive pulmonary disease (COPD) exacerbations.

ELIGIBILITY:
Main Inclusion criteria:

* Diagnosis of COPD
* Post-bronchodilator FEV1<80% predicted and FEV1/FVC<70% predicted

Main Exclusion criteria:

* Significant other diseases then COPD
* Recent myocardial infarction (MI)
* Unstable or life-threatening arrythmia requiring intervention or change in drug therapy
* Hospitalisation for cardiac failure in past year
* History of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2008-11-21 (Actual); Study Completion 2008-11-21 (Actual)

PRIMARY OUTCOMES:
Trough forced expiratory volume in one second (FEV1) response | 12 Weeks, 24 Weeks and 48 Weeks
FEV1 area under the curve (AUC) 0-8h response | 12 Weeks, 24 Weeks and 48 Weeks
Mahler Transition Dyspnoea Index (TDI) focal score | 12 Weeks, 24 Weeks and 48 Weeks
St George Respiratory Questionnaire (SGRQ) total score | 12 Weeks, 24 Weeks and 48 Weeks
Time to first moderate to severe COPD exacerbation | 12 Weeks, 24 Weeks and 48 Weeks

SECONDARY OUTCOMES:
FEV1 AUC 0-8h response | 4, 36 and 48 weeks
Trough FEV1 response | 4, 36 and 48 weeks
Peak FEV1 response | 12, 24, 36 and 48 weeks
Use of rescue medication (weekly mean number of puffs of as-needed salbutamol/albuterol per day, daytime and night-time) | 24 hours
Forced vital capacity (FVC) AUC0-8h and trough FVC response | 48 weeks
Individual FEV1, FVC and peak expiratory flow (PEF) measurements | 48 weeks
Weekly mean morning pre-dose and evening pre-dose PEFs and FEV1 (recorded by Asthma Monitor® 2 (AM2+)); PEFs determined by spirometry ] | 48 weeks
Weekly mean number of COPD related night time awakenings | 1 week
Mahler TDI focal score | 4, 36 and 48 weeks
Mahler Dyspnoea Indices (Functional Impairment, Magnitude of Task and Magnitude of Effort) | 4, 12, 24, 36 and 48 weeks
SGRQ total score, and the impact, activity and symptoms domain scores from the SGRQ | 4, 12, 36 and 48 weeks
All adverse events | 48 weeks
Vital signs: pulse rate and blood pressure | Baseline and 4 weeks
Routine blood chemistry, haematology and urinalysis | Baseline and 48 weeks
Vital status of randomised patients | 48 weeks
Number of days in hospital (including ambulance transportation | 48 weeks
Number of unscheduled health care provider visits | 48 weeks
Number of visits in emergency room (including ambulance transportation) | 48 weeks
Number of days in intensive care unit | 48 weeks
Concomitant medications (for instance antibiotics and systemic steroids). | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (72):
- United States (20):
  - 1184.14.01013 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1184.14.01018 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1184.14.01006 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1184.14.01003 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1184.14.01015 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 1184.14.01007 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1184.14.01005 Boehringer Ingelheim Investigational Site, Bangor, Maine
  - 1184.14.01020 Boehringer Ingelheim Investigational Site, Edina, Minnesota
  - 1184.14.01009 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1184.14.01002 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1184.14.01021 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1184.14.01012 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1184.14.01017 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1184.14.01008 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1184.14.01014 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1184.14.01022 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1184.14.01001 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1184.14.01010 Boehringer Ingelheim Investigational Site, Temple, Texas
  - 1184.14.01011 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1184.14.01019 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- 1184.14.43001 Boehringer Ingelheim Investigational Site, Feldbach, Austria
- Belgium (2):
  - 1184.14.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1184.14.32004 Boehringer Ingelheim Investigational Site, Turnhout
- Canada (7):
  - 1184.14.02005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1184.14.02003 Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - 1184.14.02010 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1184.14.02001 Boehringer Ingelheim Investigational Site, Niagara Falls, Ontario
  - 1184.14.02002 Boehringer Ingelheim Investigational Site, La Malbaie, Quebec
  - 1184.14.02008 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
  - 1184.14.02007 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Denmark (2):
  - 1184.14.45001 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1184.14.45002 Boehringer Ingelheim Investigational Site, København NV
- Estonia (2):
  - 1184.14.37202 Boehringer Ingelheim Investigational Site, Tallinn
  - 1184.14.37201 Boehringer Ingelheim Investigational Site, Tartu
- Finland (2):
  - 1184.14.35802 Boehringer Ingelheim Investigational Site, Espoo
  - 1184.14.35801 Boehringer Ingelheim Investigational Site, HUS
- France (6):
  - 1184.14.3301A Boehringer Ingelheim Investigational Site, Brest
  - 1184.14.3304A Boehringer Ingelheim Investigational Site, Marseille
  - 1184.14.3302A Boehringer Ingelheim Investigational Site, Montpellier
  - 1184.14.3303A Boehringer Ingelheim Investigational Site, Perpignan
  - 1184.14.3303B Boehringer Ingelheim Investigational Site, Perpignan
  - 1184.14.3303C Boehringer Ingelheim Investigational Site, Perpignan
- Germany (7):
  - 1184.14.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.14.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.14.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.14.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 1184.14.49002 Boehringer Ingelheim Investigational Site, Hamburg
  - 1184.14.49007 Boehringer Ingelheim Investigational Site, Hamburg
  - 1184.14.49001 Boehringer Ingelheim Investigational Site, Leipzig
- Greece (3):
  - 1184.14.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1184.14.30004 Boehringer Ingelheim Investigational Site, Nafplion
  - 1184.14.30006 Boehringer Ingelheim Investigational Site, Rethymno
- Hungary (4):
  - 1184.14.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 1184.14.36001 Boehringer Ingelheim Investigational Site, Hodmezövasarhely
  - 1184.14.36005 Boehringer Ingelheim Investigational Site, Komló
  - 1184.14.36004 Boehringer Ingelheim Investigational Site, Miskolc
- 1184.14.39001 Boehringer Ingelheim Investigational Site, Pisa, Italy
- Latvia (3):
  - 1184.14.37101 Boehringer Ingelheim Investigational Site, Krāslava
  - 1184.14.37103 Boehringer Ingelheim Investigational Site, Kuldīga
  - 1184.14.37102 Boehringer Ingelheim Investigational Site, Talsi
- 1184.14.37003 Boehringer Ingelheim Investigational Site, Klaipėda, Lithuania
- Netherlands (4):
  - 1184.14.31004 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1184.14.31003 Boehringer Ingelheim Investigational Site, Heerlen
  - 1184.14.31002 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 1184.14.31001 Boehringer Ingelheim Investigational Site, Veldhoven
- 1184.14.42103 Boehringer Ingelheim Investigational Site, Bardejov, Slovakia
- South Korea (3):
  - 1184.14.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1184.14.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1184.14.82003 Boehringer Ingelheim Investigational Site, Seoul
- Sweden (3):
  - 1184.14.46002 Boehringer Ingelheim Investigational Site, Linköping
  - 1184.14.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1184.14.46003 Boehringer Ingelheim Investigational Site, Sundsvall

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/